CLINICAL TRIAL: NCT05978206
Title: Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Nandrolone Decanoate Therapy and Therapy With Complex Physiotherapy and Diet in the Treatment of Sarcopenia
Brief Title: Study of the Effectiveness of Treatment of Sarcopenia With the Use of a Medicinal Product (Nandrolone), Comprehensive Physiotherapy and Diet
Acronym: SARKOPENIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIGRIR_002SARKOPENIA
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Nandrolone Decanoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nandrolone (Experimental)
  Interventions: Drug: Nandrolone Decanoate; Behavioral: Physiotherapy Intervention; Behavioral: Nutritional Intervention
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Physiotherapy Intervention; Behavioral: Nutritional Intervention; Drug: Placebo

INTERVENTIONS:
Drug: Nandrolone Decanoate — Patients will receive nandrolone decanoate (1 ml, 50 mg/ml intramuscularly given per visit) or placebo
  Arms: Nandrolone
Behavioral: Physiotherapy Intervention — The physiotherapeutic intervention includes the following components:
  1. Strength training will include strength exercises 3 x a week x 30 min - load from 60% to 80% 1RM for individual muscle groups, - 10 repetitions of the exercise, - 1-3 series in 1 session (break between sessions 60 seconds).
  2. Endurance training will include aerobic exercises (cycle ergometer, treadmill, general fitness exercises) 3 times a week x 30 minutes, load from 60% to 80% of maximum heart rate.
Behavioral: Nutritional Intervention — An individual diet in terms of calorific value and the content of energy substrates - proteins, fats and carbohydrates, as well as other nutrients, in accordance with specific nutrition standards.
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a single-center, prospective, randomized, double-blind (pharmacotherapy), placebo-controlled, and comprehensive physiotherapy and nutritional intervention phase II clinical trial to determine the usefulness of nandrolone decanoate in a new indication (sarcopenia).

Patients will be randomized 1:1 to receive nandrolone decanoate (50 mg intramuscular injection over four visits every 3 weeks) or placebo (1 ml volume equivalent to 50 mg intramuscular nandrolone decanoate dose) for 12 weeks (83-85 days ). Both groups will receive comprehensive physiotherapy and nutritional intervention.

There will be 5 outpatient visits to the research center. The procedures and assessments performed as part of the study are listed in the study schedule.

It is planned to include 168 patients in the study, which, assuming a 10% level of non-completion of the program, will result in the examination of 152 patients (76 in each arm). The study will cover people aged over 60 to 99 years of age with confirmed muscle weakness measured with a hand dynamometer (< 27 kg for men and 16 kg for women) and with a decrease in: muscle mass of upper and lower limbs (ASMM) (7.0 kg/m2 height in men and 5.5 kg/m2 in women) or total muscle mass of the upper and lower extremities (< 20 kg in men and < 15 kg in women) by densitometry.

ELIGIBILITY:
Inclusion Criteria:

1. individuals aged 60 years or older through 99 years of age.
2. Patients meeting the following criteria diagnosed with sarcopenia based on EWGSOP 2 criteria from 2019:

   * weakness of muscle strength measured by hand dynamometer ( < 27 kg for men and 16 kg for women) and
   * reduction in densitometry:

     * upper and lower limb muscle mass (ASMM)(below 7.0 kg/m2 height in men and 5.5 kg/m2 in women) or
     * total muscle mass of the arms and legs in men less than 20 kg and less than 15 kg in women).

Exclusion Criteria:

1. Mini-Mental State Examination (MMSE) score less than 24;
2. malignant neoplasm, lymphoproliferative or myeloproliferative disorders requiring oncologic or palliative treatment and the period before: 5 years in the case of: malignant melanoma, leukemia, Hodgkin's disease, malignant lymphomas, kidney tumors, 12 months in the case of other malignant neoplasms after the completion of surgery, chemotherapy or radiotherapy;
3. history of oncologic diagnosis of focal lesions in the prostate gland;
4. acute and chronic inflammatory diseases of the gastrointestinal tract that present with malabsorption (celiac disease, ulcerative colitis, Crohn's disease, etc.);
5. uncompensated hyper- or hypothyroidism;
6. recent history of myocardial infarction or stroke (up to 4 weeks prior to study entry); history of thromboembolism (up to 6 months prior to study entry) or recurrent thromboembolism;
7. poorly controlled hypertension;
8. liver impairment (AST and/or ALT > 3x normal: AST> 111 U/l and ALT> 123 U/l); 9 Acute kidney injury and/or chronic kidney disease (stage G4 and G5);

10. nephrotic syndrome, acute or chronic glomerulonephritis; 11. advanced circulatory failure (NYHA stages III and IV); 12. Acute and chronic respiratory failure requiring oxygen therapy; 13. Amyotrophic lateral sclerosis, multiple sclerosis, myasthenia gravis, dystrophies, spinal muscular atrophy type IV, primary muscular disorders (ICD-10 G71), toxic-field myopathies, myopathies in the course of infectious and parasitic diseases. Epilepsy; 14. need for treatment during the study period:

* systemic corticosteroids for more than 3 weeks at a dose equivalent to greater than or equal to 5 mg prednisone;
* hormone replacement therapy,
* 5-alpha reductase inhibitors,
* aromatase inhibitors,
* anti-estrogenic hormonal drugs with anabolic effects other than nandrolone decanoate,
* megestrol. 15. Lack of informed consent for participation in the study.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in physical fitness as assessed by the SPPB test score | in the 12th week of the study
  Change in physical fitness as assessed by the SPPB test score (4- meter gait speed test version) in points, at the 5th study visit relative to the test score performed at visit 1
Change in the 400-meter walk test score | in the 12th week of the study
  Change in the 400-meter walk test score in time units, at the 5th test visit, relative to the test score taken at visit 1

SECONDARY OUTCOMES:
lower limb muscle strength | in the 6th and 12th week of the study
  lower limb muscle strength assessed with the result of the test of getting up 5 times from a chair per unit of time, upper limb muscle strength assessed with the result of the dynamometric handgrip test in kilograms during the 3rd and 5th visit of the examination in relation to the result made during the 1st visit
Respiratory muscle strength | in the 6th and 12th week of the study
  Respiratory muscle strength assessed as a result of changes in airway pressures during inhalation and exhalation during the 5th visit of the study in relation to the result of the test performed at visit 1
muscle mass | in the 6th and 12th week of the study
  muscle mass: assessed on the basis of the content of lean body mass of the upper and lower limbs in the study of body composition analysis using the electrical bioimpedance method; during the 3rd and 5th study visit in relation to the result of the study performed during visit 1
muscle mass of the upper and lower limbs | in the 6th and 12th week of the study
  muscle mass of the upper and lower limbs: assessed on the basis of the content of lean body mass of the upper and lower limbs in the densitometry test during the 5th visit of the study in relation to the result of the test performed during visit 1
score of the Sarc-QoL quality of life questionnaire (validated Polish version) | in the 6th and 12th week of the study
  score of the Sarc-QoL quality of life questionnaire (validated Polish version) during the 5th visit of the study in relation to the result of the study performed during visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Targowski, Prof. PhD, MD, Principal Investigator — National Institute of Geriatrics, Rheumatology and Rehabilitation
Locations (1):
- Centrum Wsparcia Badań Klinicznych, Warsaw, Masovian Voivodeship, Poland